CLINICAL TRIAL: NCT03619954
Title: A Clinical Research of Natural Killer (NK) Cells Infusion for the Treatment of Advanced Malignant Tumor
Brief Title: NK Cells Infusion for Advanced Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Yue-Yin Pan, Professor of Department of Medical Oncology, Anhui Provincial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHP2018070101
Record Dates: First submitted 2018-07-06; First posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Immunotherapy
Keywords: NK cell infusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NK cells infusion (Experimental)
  Interventions: Biological: NK cells infusion

INTERVENTIONS:
Biological: NK cells infusion — Pretreatment：patients enrolled in this study will receive 20 mg/kg of cyclophosphamide for solid tumor or 20-60 mg/kg of cyclophosphamide for hematological tumor once daily for 3 times. NK cells infusion is allowed within 2-14 days after treatment.
  NK cells infusion：30-60 minutes before infusion，ant-allergic agents are applied (promethazine 25mg,i.m. ; Cimetidine 0.4g i.v. ; diphenhydramine 50mg po.). NK cells are intravenously infused into patients with 15-30 minutes every other day for one to three times. The number of every infused NK cells is 1-3×10^7/kg, counted as the number of CD56+ cells. Patients with severe pleural or ascites can also receive pleural or abdominal cavity perfusion simultaneously. The total number of infused NK cells is no more than 5×10^9 cells. 4 hours after NK cells infusion，IL-2 is applied every other day for six times

SUMMARY:
This study is designed to explore the safety and efficacy of natural killer (NK) cell infusion as treatment for patients with advanced malignant tumors after multiline therapy, and to evaluate the pharmacokinetics of NK cells in patients

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced malignant tumors diagnosed by pathological histology and/or cytology who have failed multi-line therapy and have no standard treatment method are unable to undergo surgery, radiation therapy, or chemotherapy;
2. Age 18-75 years old (≥18, ≤75);
3. ECOG: 0-1;
4. Priority should be given to the inclusion of ovarian cancer, malignant leukemia, lymphoma, etc. that have been shown to respond well to NK cell therapy;
5. Expected survival period ≥ 3 months;
6. Hematology tests also meet the following requirements:

1) WBC≥3×109/L, ANC≥1.5×109/L, Hb≥90g/L, PLT≥100×109/L; 2) TBIL ≤ 1.5 × ULN (normal upper limit), ALT and AST ≤ 2 × ULN (if there is liver metastasis, then ≤ 5 × ULN); 3) Endogenous creatinine clearance ≥ 60 ml/min (calculated based on Cockcroft-Gault formula); (7) Length of solid tumors do not exceed 6 cm; (8) Signing of informed consent from each patient

Exclusion Criteria:

1. History of other malignancies with a disease-free period <5 years (except for cured basal cell carcinoma of the skin, cured carcinoma of the cervix in situ, and gastrointestinal tumors proven to be cured by endoscopic mucosal resection);
2. Patients with brain metastases (unless the investigator believes that brain metastasis is currently stable, it is generally not recommended for enrollment);
3. Transplant recipients;
4. T-cell lymphoma patients;
5. Allergies to biologics used in this treatment;
6. Patients with HIV and syphilis;
7. HBV carriers;
8. Patients who are undergoing radiation therapy or immunotherapy within 4 weeks;
9. Patients who have undergone high-dose radiation therapy on the lung and liver within 4 months;
10. Patients with pulmonary inflammation determined by chest radiography;
11. Oxygen saturation ≤ 90% on room air;
12. Patients with cachexia caused by advanced tumors;
13. Long-term use of immunosuppressive drugs or patients who are using immunosuppressive drugs;
14. Those with serious autoimmune diseases;
15. Patients with organ failure (grade 4 of heart function; liver function with Child class C or above; brain metastasis with disturbance of consciousness; severe respiratory failure symptoms);
16. Active infections (including intra-abdominal infections).
17. Researchers consider it inappropriate to participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Successful expansion of NK cells in patient's circulatory system | 7 days after the last treatment
  CD56 positive cells ≥100 cells/μL in blood is considered as successful expansion of NK cells
Objective Response Rate | 4 weeks after all the treatment finished
  The percentage of patients who reach complete response（CR）or partial response （PR）after all treatment finished. The response is evaluated according to irRECIST.

SECONDARY OUTCOMES:
Overall survival | 1 and 2 years after treatment
  The interval time from the date when patients are enrolled into study to death or the last visit
Disease progression free survival | 1 and 2 years after treatment
  The interval time from the date when patients are enrolled into study to disease progression, death or last visit
Dynamic changes of NK cells number in blood | Day 1,3,5,7,10,14,21,28 and 2, 3, 6 months after NK cells infusion finished
  Numbers of CD56 positive cell in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Yueyin Pan, PhD, Principal Investigator — Anhui Province Cancer Center
Locations (1):
- Anhui Provincial cancer center, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided